CLINICAL TRIAL: NCT02980679
Title: A Pivotal Phase III Study of Cyclotron-produced Tc-99m Pertechnetate (CTC) Compared to Generator-produced Tc-99m Pertechnetate (G-PERT) in Subjects With Thyroid Disorders
Brief Title: A Study to Compare the Safety and Imaging Pattern of Cyclotron-produced Technetium (CTC) vs. Generator-produced Technetium (G-PERT) in People With Thyroid Disorders Who Need Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DX-CTC-003; HREBA.CC-16-0695 (Other: Health Research Ethics Board of Alberta Cancer Committee)
Record Dates: First submitted 2016-11-22; First posted 2016-12-02 (Estimated); Last update posted 2022-04-11 (Actual); Status verified 2018-11

CONDITIONS: Thyroid Gland Diseases
MeSH Terms: conditions — Thyroid Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CTC and G-PERT Imaging (Experimental): One experimental (CTC) and one standard (G-PERT) scan, at least 48 hours apart, before thyroid surgery. The order of the scans will be randomized.
  Interventions: Drug: CTC; Drug: G-PERT

INTERVENTIONS:
Drug: CTC — After injection of CTC, a whole body and thyroid scan will be performed.
  Other Names: Cyclotron-produced technetium
Drug: G-PERT — After injection of G-PERT, a whole body and thyroid scan will be performed.
  Other Names: Generator-produced technetium

SUMMARY:
A 99mTc Pertechnetate (G-PERT) scan is a nuclear medicine test that can create an image of the thyroid gland and other organs. G-PERT is approved by Health Canada for the direct imaging and measurement of thyroid uptake.

Doctors and researchers at the University of Alberta have developed a new method of producing 99mTc Pertechnetate (called CTC). It is made in a cyclotron at the Medical Isotope and Cyclotron Facility (MICF) at the University of Alberta, Edmonton, Alberta. This new production method will provide another source of 99mTc Pertechnetate. The aim of this study is to confirm that CTC is safe and can be used interchangeably with G-PERT.

DETAILED DESCRIPTION:
The clinical trial will be a Phase III, prospective, crossover, image interpretation blinded, single site study. All subjects will receive Tc-99m pertechnetate (one CTC and one G-PERT administration separated by at least 48 hours) and subsequently be imaged for thyroid uptake and whole body biodistribution. The order of the scans will be randomized. The thyroid image will be interpreted for uptake / no uptake in the thyroid, and the whole body biodistribution image will be interpreted for uptake / no uptake in selected anatomical sites. Interpretation of thyroid imaging results will be compared with other clinical findings (such as pre-surgical ultrasound, fine needle aspirate, and post-surgical pathology results, when available). All imaging assessments will be conducted by 1 blinded Nuclear Medicine physician. A safety evaluation will be conducted on all subjects receiving CTC, consisting of vital signs, haematology and SMA-12 serum biochemistry profile (pre-injection and post-imaging), and, for both CTC and G-PERT, an adverse event assessment (until the subject leaves the Nuclear Medicine department) after each administration.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 18 years of age and < 80 years of age.
2. Have a proven or suspected thyroid pathology that requires surgery by standard clinical criteria.
3. Able and willing to follow instructions and comply with the protocol.
4. Provide written informed consent prior to participation in the study.

Exclusion Criteria:

1. Nursing or pregnant females.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-03-03 (Actual); Primary Completion 2019-02-25 (Actual); Study Completion 2019-02-25 (Actual)

PRIMARY OUTCOMES:
Clinical Comparability of CTC with G-PERT | up to 1 year
  The primary efficacy endpoint is the clinical comparability of CTC with G-PERT consisting of a combination of the following results:
  1. A thyroid image, assessed for uptake or no uptake in the thyroid.
  2. A whole body biodistribution study, assessed for uptake or no uptake in selected anatomical areas.

SECONDARY OUTCOMES:
Change in vital signs after CTC injection | Before CTC injection and after CTC scan (within ~30 min)
  Vital signs are measured before injection of CTC and after CTC scan and changes will be summarized.
Changes in haematology / SMA-12 serum biochemistry after CTC injection | Before CTC injection and after CTC scan (within ~30 min)
  A blood sample is drawn before injection of CTC and after CTC scan. The haematology and SMA-12 serum biochemistry parameters will be recorded and all changes will be summarized.
Number of participants with adverse events | up to 1 year
  Subjects will be monitored for adverse events after CTC and G-PERT scans while in the Nuclear Medicine Department. All adverse events observed or reported will be recorded and assessed.
Correlation of CTC with other clinical findings | up to 1 year
  Correlation of thyroid images with other clinical findings (such as pre-surgical ultrasound, FNA, and post-surgical pathology results, when available).
CTC diagnostic outcomes and parameters | up to 1 year
  Calculation of diagnostic outcomes (TP, TN, FP, FN) and the corresponding diagnostic parameters (sensitivity, specificity, accuracy).
Overall clinical comparability of CTC with G-PERT | up to 1 year
  The overall clinical comparability of CTC with G-PERT using diagnostic outcomes (True Positive, True Negative, False Positive, False Negative) to determine the corresponding diagnostic parameters (sensitivity, specificity, accuracy).

CONTACTS AND LOCATIONS:
Overall Officials: Todd P McMullen, MD, PhD, FRCSC, FACS, Principal Investigator — Associate Professor of Surgery and Oncology; Director, Division of Surgical Oncology, Department of Oncology
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No